CLINICAL TRIAL: NCT07268690
Title: Risk-Adapted Omission of Level Va Irradiation in Nasopharyngeal Carcinoma: A Phase III Randomized Non-Inferiority Trial
Brief Title: Risk-Adapted Omission of Level Va Irradiation in Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPC013
Record Dates: First submitted 2025-11-23; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Nasopharyngeal Carcinoma by AJCC V9 Stage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- level Va-sparing IMRT (Experimental): Level Va irradiation is omitted except in the presence of any of the following high-risk features:
  1. Ipsilateral Level IIb involvement;
  2. Ipsilateral Level III nodes involvement;
  3. Ipsilateral positive lymph nodes below the cricoid cartilage (Level IV or Vb-c);
  Interventions: Radiation: Omission of Level Va Irradiation in Nasopharyngeal Carcinoma
- level Va-covering IMRT (No Intervention): Level Va is routinely irradiated according to CACA/CMDA guidelines.

INTERVENTIONS:
Radiation: Omission of Level Va Irradiation in Nasopharyngeal Carcinoma — Level Va should be irradiated only in the presence of any of the following high-risk features: 1. Ipsilateral Level IIb involvement; 2. Ipsilateral Level III nodes involvement; 3. Ipsilateral positive lymph nodes below the cricoid cartilage (Level IV or Vb-c).
  Arms: level Va-sparing IMRT

SUMMARY:
This is a randomized, phase III, prospective, multi-center trial in newly diagnosed nasopharyngeal carcinoma (NPC) patients without distant metastasis. This study will evaluate whether omitting Level Va irradiation in patients without these risk features does not compromise regional control or survival, with the goal of providing robust evidence to guide further personalization of NPC radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologic diagnosis (pathologically confirmed by nasopharyngeal biopsy) was nasopharyngeal carcinoma;
2. No distant metastatic;
3. Eastern Cooperative Oncology Group (ECOG) score of 0 or 1;
4. Signing informed consent;
5. Follow up regularly and comply with test requirements.

Exclusion Criteria:

1. Ipsilateral Level IIb involvement;
2. Ipsilateral Level III nodes involvement;
3. Ipsilateral positive lymph nodes below the cricoid cartilage (Level IV or Vb-c);
4. Disease progression during IMRT;
5. Previous malignancy or other concomitant malignant diseases;
6. The evaluation information of tumor efficacy can not be obtained;
7. Receive blind treatment in other clinical research;
8. Have or are suffering from other malignant tumors within 5 years (except non- melanoma skin cancer or pre-invasive cervical cancer);
9. Serious complications, such as uncontrolled hypertension, coronary heart disease, diabetes, heart failure, etc;
10. Active systemic infection;
11. No or limited capacity for civil conduct;
12. The patient has a physical or mental disorder, and the researcher considers that the patient is unable to fully or fully understand the possible complications of this study;
13. Pregnancy or lactation period;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Regional failure-free survival | 3 years
  The regional relapse-free survival rate will be estimated using Kaplan-Meier method for each arm from the date of randomization to the date of nodal relapse or death from any cause, whichever occurred first. Their differences will be compared between treatment arms using the log-rank test.

SECONDARY OUTCOMES:
overall survival | 3 years
  time from the date of the start of chemotherapy to death due to any cause
Distant metastasis-free survival | 3 years
  The distant metastasis-free survival rate will be estimated using Kaplan-Meier
Local failure-free survival | 3 years
  until documented treatment local failure or death from any cause.
Patient's quality-of-life | 3 years
  European Organization for Research and Treatment of Cancer Quality-of-Life Head and Neck Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Qiaojuan Guo, Study Chair — Fujian Cancer Hospital
Locations (1):
- Fujian Cancer hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No